CLINICAL TRIAL: NCT03988504
Title: Impact of Predictive Genetic Testing on Quality of Life and Health-related Behaviour
Brief Title: Impact of Predictive Genetic Testing
Status: Completed | Type: Observational
Sponsor: Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Mark Dominik Alscher, Medical Director, Managing Director, Robert Bosch Medical Center
Other Study IDs: RBK 358
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Genetic Testing; Quality of Life; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Routine check up including genetic testing — Intervention is a routine check up including preemptive genetic testing

SUMMARY:
Analysing Impact of preemptive genetic testing on quality of life, physical activity and eating behavior at baseline and 3 months after testing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* informed consent for genetic testing
* informed consent for study participation

Exclusion Criteria:

* Age <18 years
* renal replacement dependency
* pregnancy
* active cancer disease
* no informed consent for genetic testing or study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects with request for health check up at Robert-Bosch-Hospital
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life assessed by the SF-36 questionnaire [followed by its scale information in the Description] | 3 months
  Short form (36) (SF-36) questionnaire evaluates health related quality of life (Scale 0-100)
Physical activity assessed by the IPAQ questionnaire [followed by its scale information in the Description] | 3 months
  International Physical Activity Questionnaire (IPAQ) evaluates physical activity in MET(metabolic equivalent)/min/week
Eating behavior assessed by the modified LEI questionnaire [followed by its scale information in the Description] | 3 months
  The modified Luzerner Ernaehrungs Index (LEI) questionnaire evaluates eating behavior at lunch (Scale 1-4 per item; 1=never; 4=daily)

SECONDARY OUTCOMES:
Satisfaction with check up and genetic testing: Likert scale (1-10) | 3 months
  Likert scale (1-10)

IPD SHARING:
Plan to Share IPD: Undecided
On request